CLINICAL TRIAL: NCT03391804
Title: Pilot Study of ALLN-177 in Adult and Pediatric Subjects Aged 12 Years or Older With Enteric or Primary Hyperoxaluria and Hyperoxalemia
Brief Title: Study of ALLN-177 in Patients Aged 12 Years or Older With Enteric or Primary Hyperoxaluria and Hyperoxalemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLN-177-206; 2017-003547-38 (EudraCT Number)
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-02

CONDITIONS: Enteric Hyperoxaluria; Primary Hyperoxaluria; Hyperoxalemia
Keywords: Oxalate; Kidney Stones; oxalate nephropathy; systemic oxalosis
MeSH Terms: conditions — Hyperoxaluria, Primary; Kidney Calculi | interventions — reloxaliase; oxalate decarboxylase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALLN-177 (Experimental): ALLN-177 7,500 units (2 capsules)
  Interventions: Drug: ALLN-177

INTERVENTIONS:
Drug: ALLN-177 — ALLN-177 7,500 units (2 capsules) with each meal/snack by mouth 5 times per day for 12 weeks
  Other Names: Oxalate decarboxylase

SUMMARY:
Evaluate the efficacy and safety of ALLN-177 in reducing plasma and urinary oxalate levels in adult and pediatric patients with enteric hyperoxaluria and hyperoxalemia or primary hyperoxaluria

DETAILED DESCRIPTION:
Phase 2, multi-center, open label, single arm study to evaluate the effect and safety of ALLN-177 in adult and pediatric patients aged 12 and older with enteric hyperoxaluria and hyperoxalemia or primary hyperoxaluria .

Approximately 15-20 evaluable subjects are planned to be enrolled in the study. Eligible subjects will administer ALLN-177 with each meal/snack 5 times per day for 12 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed a informed consent form or an assent
2. Aged 12 or older with body weight ≥ 35kg
3. History of primary hyperoxaluria or enteric hyperoxaluria associated with a known underlying enteric disorder associated with malabsorption (e.g., bariatric surgery, Crohn's disease, short bowel syndrome, or other malabsorption syndrome)
4. Urinary oxalate ≥ 40mg/24h (normalized for body surface area in children) at Screening in patients with eGFR >15 mL/min/1.73m2
5. In patients with enteric hyperoxaluria, eGFR < 45mL/min/1.73m2 at Screening
6. In patients with enteric hyperoxaluria, plasma oxalate > 5µmol/L at Screening
7. Patients on dialysis, must be stable for greater than 3 months

Exclusion Criteria:

1. Unable or unwilling to discontinue Vitamin C supplementation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Change in plasma oxalate | on 12 weeks of treatment
  Efficacy will be assessed based on change from baseline in plasma oxalate

SECONDARY OUTCOMES:
Change in 24-hr urinary oxalate excretion | on 12 weeks of treatment
  Efficacy will be assessed based on change from baseline in 24-hr urinary oxalate excretion

CONTACTS AND LOCATIONS:
Overall Officials: David Clark, MD, Study Director — Allena Pharmaceuticals Inc
Locations (9):
- United States (4):
  - Mayo Clinic, Scottsdale, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Yale University School of Medicine, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota
- Charite Campus Berlin-Mitte, Medizinische Klinik mit Schwepunkt Nephrologie und Internistische Intensivmedizin, Berlin, Germany
- United Kingdom (4):
  - Wellcome Trust Clinical Research Facility, Southampton, Hampshire
  - Royal Preston Hospital, Preston, Lancashire
  - Leeds General Infirmary, Leeds
  - Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No